CLINICAL TRIAL: NCT00005264
Title: Pediatric Epidemiology of Cardiovascular Disease Risk Factors (Project Heartbeat)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1148; U01HL041166 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2002-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Atherosclerosis

SUMMARY:
To conduct a longitudinal, natural history study of cardiovascular disease risk factors in children. Growth curves were compared for levels of blood pressure, lipids, cardiac structures and function, and related to physical growth and maturation, nutrient intake, physical activity, body composition, puberty, and smoking.

DETAILED DESCRIPTION:
BACKGROUND:

Both the pathologic precursors of atherosclerosis and the development of its major risk factors -- blood pressure, blood lipids, and cigarette smoking -- are often far advanced before age 20 or within the period from birth or conception through adolescence. In 1990, there was growing interest in understanding these aspects of human biology and in devising appropriate preventive measures.

In 1990, knowledge about the risk factors during childhood and adolescence was based mainly on cross-sectional surveys, from which very striking and consistent patterns of change with age were inferred, and from which reference values for screening and management were derived. Both growth and sexual maturation influence these patterns strongly, yet these risk factors had only recently been taken into account in 1990, only partially in screening recommendations for blood pressure and not at all for cholesterol.

DESIGN NARRATIVE:

Subjects were selected by simple random sampling. Data were collected on dependent variables including blood pressure, heart rate, echocardiography, Doppler flow, blood lipids, and smoking. Independent variables included growth, diet and nutrition, electrolytes, physical activity and fitness, personal, family, and social history, and bone age. Most observations were recorded at four month intervals. There was a six month pretest recruitment period, four years of cycled measurements and data collection, and six months of analysis and reporting. Curves for both velocity and acceleration of growth for attained levels of blood pressure, blood lipids, and smoking were determined as were longitudinal relationships between individual growth curves of blood pressure, echocardiographic measures, physical growth, sexual maturation, body composition, diet, physical activity, and social factors.

Dr. Labarthe has several R03 grants to analyze data from Project Heartbeat. See also Study 4962.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-09; Study Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darwin LaBarthe — University of Texas

REFERENCES:
- [Background] Tanner JM, Oshman D, Lindgren G, Grunbaum JA, Elsouki R, Labarthe D. Reliability and validity of computer-assisted estimates of Tanner-Whitehouse skeletal maturity (CASAS): comparison with the manual method. Horm Res. 1994;42(6):288-94. doi: 10.1159/000184211. PMID 7698726
- [Background] Labarthe DR, Nichaman MZ, Harrist RB, Grunbaum JA, Dai S. Development of cardiovascular risk factors from ages 8 to 18 in Project HeartBeat! Study design and patterns of change in plasma total cholesterol concentration. Circulation. 1997 Jun 17;95(12):2636-42. doi: 10.1161/01.cir.95.12.2636. PMID 9193432
- [Background] Grunbaum JA, Labarthe DR, Ayars C, Harrist R, Nichaman MZ. Recruitment and enrollment for Project HeartBeat! Achieving the goals of minority inclusion. Ethn Dis. 1996 Autumn;6(3-4):203-12. PMID 9086310
- [Background] Dai S, Ayres NA, Harrist RB, Bricker JT, Labarthe DR. Validity of echocardiographic measurement in an epidemiological study. Project HeartBeat! Hypertension. 1999 Aug;34(2):236-41. doi: 10.1161/01.hyp.34.2.236. PMID 10454447
- [Background] Fulton JE, Dai S, Grunbaum JA, Boerwinkle E, Labarthe DR. Apolipoprotein E affects serial changes in total and low-density lipoprotein cholesterol in adolescent girls: Project HeartBeat! Metabolism. 1999 Mar;48(3):285-90. doi: 10.1016/s0026-0495(99)90073-2. PMID 10094101
- [Background] Tanner J, Oshman D, Bahhage F, Healy M. Tanner-Whitehouse bone age reference values for North American children. J Pediatr. 1997 Jul;131(1 Pt 1):34-40. doi: 10.1016/s0022-3476(97)90000-7. PMID 9255189
- [Background] Dai S, Labarthe DR, Grunbaum JA, Harrist RB, Mueller WH. Longitudinal analysis of changes in indices of obesity from age 8 years to age 18 years. Project HeartBeat! Am J Epidemiol. 2002 Oct 15;156(8):720-9. doi: 10.1093/aje/kwf109. PMID 12370160
- [Background] Mueller WH, Harrist RB, Doyle SR, Ayars CL, Labarthe DR. Body measurement variability, fatness, and fat-free mass in children 8, 11, and 14 years of age: Project HeartBeat! Am J Hum Biol. 1999;11(1):69-78. doi: 10.1002/(SICI)1520-6300(1999)11:13.0.CO;2-T. PMID 11533935
- [Background] Mueller WH, Grunbaum JA, Labarthe DR. Anger expression, body fat, and blood pressure in adolescents: Project HeartBeat! Am J Hum Biol. 2001 Jul-Aug;13(4):531-8. doi: 10.1002/ajhb.1085. PMID 11400224